CLINICAL TRIAL: NCT00817024
Title: Clinical Study of Herbal Formula in Post PCI Patients.
Brief Title: Study of Herbal Formula Corresponding to Syndrome in Treating Post Percutaneous Coronary Intervention (PCI) Patients With Coronary Heart Disease (CHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: China Academy of Chinese Medical Sciences, Guang'an Men Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNSF90709048
Record Dates: First submitted 2009-01-04; First posted 2009-01-06 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; PCI; Traditional Chinese Medicine; Quality of Life
MeSH Terms: conditions — Coronary Disease | interventions — Xue-Fu-Zhu-Yu decoction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Xuefu Zhuyu Capsules (Experimental)
  Interventions: Drug: Xuefu Zhuyu Capsules Plus Placebo of Sheng Mai Capsules,
- Sheng Mai Capsules (Active Comparator)
  Interventions: Drug: Sheng Mai Capsules Plus Placebo of Xuefu Zhuyu Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of Xuefu Zhuyu Capsules Plus Placebo of Sheng Mai Capsules

INTERVENTIONS:
Drug: Xuefu Zhuyu Capsules Plus Placebo of Sheng Mai Capsules, — 3# XFZY capsules plus 3# placebo of SM capsules, po, Tid, for 4 weeks
  Arms: Xuefu Zhuyu Capsules
Drug: Sheng Mai Capsules Plus Placebo of Xuefu Zhuyu Capsules — 3# SM capsules plus 3# placebo of XFZY capsules, po, Tid, for 4 weeks
  Arms: Sheng Mai Capsules
Drug: Placebo of Xuefu Zhuyu Capsules Plus Placebo of Sheng Mai Capsules — 3# Placebo of XFZY capsules plus 3# placebo of SM capsules, po, Tid, for 4 weeks
  Arms: Placebo

SUMMARY:
We conduct this clinical trial to determine the effects of Xuefu Zhuyu capsule (based on TCM "Zheng Hou" theory) in helping recovery from coronary heart disease(CHD)after PCI and find out whether this kind of effecacy is much better within patients administered with TCM syndrome-based individualized medication.

DETAILED DESCRIPTION:
The effectiveness of a Chinese herbal formulae is not completely based on the disease or some biomedical indexes, but much more on the TCM syndrome(Chinese name:Zheng Hou)which is generalized from patients' TCM signs and symptoms. Thus, conventional medical curative effecacy evaluation system seems not to so fit for TCM clinical studies. Although many clinical studies from Chinese literature have reported the beneficial effects of various of TCM herbal agents in improving symptoms and signs as well as antagonism of specific pathological changes in CHD patients, most of these trials are lack of well-designed methodologies and the reliability of results still remains unclear. Therefore, we designed this clinical trial, with a randomized, placebo controlled way, to evaluate the curative effects of Xuefu Zhuyu capsule(a Chinese herbal medicine)in patients with Post-PCI CHD patients and find out whether this effects will be better displayed within subjects administered with syndrome-based individualized medication.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Clinical diagnosis of coronary heart disease (confirmed by coronary angiography)
* Successfully received interventional therapy (PTCA or PCI)
* belong to TCM blood-stasis syndrome
* Must be able to swallow tablets
* Able to give written informed consent

Exclusion Criteria:

* Symptomatic congestive heart failure(New York Heart Association class III-IV)
* Females during pregnancy or lactation
* Serious dysfunction in important organs (liver, lung, kidney，et al)
* Use of concomitant Chinese herbal medicine
* Already attend other clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Severity of anginal attacks, alternations of TCM symptoms and signs, and electrocardiographic changes. | 4 weeks

SECONDARY OUTCOMES:
Health related quality of life (Hr-QoL); Changes in serum lipid, inflammatory reaction level and endothelial function status alternations before and after the treatment. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, M.D., Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospital, Beijing, China

REFERENCES:
- [Derived] Chu FY, Wang J, Yao KW, Li ZZ. Effect of Xuefu Zhuyu Capsule (血府逐瘀胶囊) on the symptoms and signs and health-related quality of life in the unstable angina patients with blood-stasis syndrome after percutaneous coronary intervention: A Randomized controlled trial. Chin J Integr Med. 2010 Oct;16(5):399-405. doi: 10.1007/s11655-010-9999-9. Epub 2010 Jun 10. PMID 20535581
- [Derived] Chu FY, Wang J, Sun XW, Xing YW, Yao KW, Wang SH, Li ZZ. [A randomized double-blinded controlled trial of Xuefu Zhuyu Capsule on short-term quality of life in unstable anginal patients with blood-stasis syndrome after percutaneous coronary intervention]. Zhong Xi Yi Jie He Xue Bao. 2009 Aug;7(8):729-35. doi: 10.3736/jcim20090805. Chinese. PMID 19671410